CLINICAL TRIAL: NCT06031844
Title: A Randomized, Placebo-controlled, Parallel-group, Investigator- and Participant-blinded Phase 2a Study to Investigate the Efficacy, Safety, and Tolerability of DFV890 for Inflammatory Marker Reduction in Adult Participants With Coronary Heart Disease and Elevated hsCRP
Brief Title: A Study to Investigate the Efficacy, Safety, and Tolerability of DFV890 for Inflammatory Marker Reduction in Adult Participants With Coronary Heart Disease and Elevated hsCRP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDFV890F12201
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Coronary Heart Disease
Keywords: DFV890; Phase 2a; coronary heart disease; elevated hsCRP
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence 1 (Experimental): Participants will be administered Placebo and different doses of DFV890
  Interventions: Drug: DFV890; Drug: Placebo
- Treatment sequence 2 (Experimental): Participants will be administered Placebo and different doses of DFV890
  Interventions: Drug: DFV890; Drug: Placebo
- Treatment sequence 3 (Experimental): Participants will be administered different doses of DFV890
  Interventions: Drug: DFV890
- Treatment sequence 4 (Placebo Comparator): Participants will be administered Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DFV890 — oral film-coated tablets
  Arms: Treatment Sequence 1; Treatment sequence 2; Treatment sequence 3
Drug: Placebo — oral film-coated tablets
  Arms: Treatment Sequence 1; Treatment sequence 2; Treatment sequence 4

SUMMARY:
This Phase 2a clinical trial will evaluate the effectiveness, safety, and tolerability of increasing dose strengths of an oral daily medication, DFV890, administered for 12 weeks, to reduce key markers of inflammation related to CVD risk, such as IL-6 and IL-18, in approximately 24 people with known heart disease and an elevated marker of inflammation, hsCRP.

DETAILED DESCRIPTION:
This is a multi-center, randomized, placebo-controlled, participant- and investigator-blinded study to evaluate the efficacy, safety, and tolerability of intra-individual dose escalation of DFV890 for inflammatory marker reduction in participants with coronary heart disease and elevated hsCRP. The study consists of a screening period of up to 60 days, a treatment period of approximately 12 weeks, an end of treatment (EOT) visit on Day 85, which is one day after the last dose on Day 84, a follow-up period of approximately 1 week and a standard safety-follow-up call approximately 30 days following the last dose. The overall study duration is approximately 24 weeks and approximately 24 participants will be enrolled into the trial.

Participants meeting all eligibility criteria will be randomized in a 5:5:1:1 ratio to one of four treatment sequences (three DFV890 treatment sequences or a placebo-only sequence). The dose of DFV890 will be uptitrated (according to the specific treatment sequence that the participant is assigned to) approximately every three weeks at the scheduled visits on Days 22, 43 and 64.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged between 18 - 85 years (inclusive) at the start of screening will be included.
* Subjects must have a body mass index (BMI) within the range of 18 - 45 kg/m2. BMI = Body weight (kg) / [Height (m)]2
* Documented spontaneous myocardial infarction (MI) (diagnosed according to the universal MI criteria with or without evidence of ST segment elevation) at least 30 days before the start of screening.
* Participants must have hsCRP levels ≥ 2 mg/L at two timepoints during screening. Screening values must be separated by a minimum of 8 days. The initial hsCRP value must be a minimum of 30 days after the qualifying MI or after any percutaneous coronary intervention (PCI) performed separately from the qualifying MI.
* For participants on statin therapy (HMG-CoA reductase inhibitor), as clinically indicated, participants must be on a stable regimen (at least 4 weeks before randomization), with no planned statin dose changes over the course of the trial treatment period. Unplanned statin dose changes during the trial treatment period may occur.

Exclusion Criteria:

* Patients receiving concomitant medications that are known to be strong or moderate inducers of cytochrome CYP2C9 enzyme and/or strong inducers of CYP3A, strong inhibitors of CYP2C9 and/or strong or moderate inhibitors of CYP3A and the treatment cannot be discontinued or switched to a different medication within 5 half-lives or 1 week (whichever is longer) prior to Day 1 and for the duration of the study.
* Patients with suspected or proven immunocompromised state at screening
* History of ongoing, chronic, or major recurrent infectious disease, at the discretion of the investigator, at the start of screening.
* Use of any biologic drugs targeting the immune system within 26 weeks of Day 1
* Multi-vessel Coronary Artery Bypass Graft (CABG) surgery within the past 6 months prior to the start of screening.
* Symptomatic Class IV heart failure (New York Heart Association) at the start of screening.
* Planned coronary revascularization (PCI or CABG) or any other major surgical procedure during the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Serum levels of IL-6 and IL-18 | From Day 22 to End of Study Visit (up to 92 days)
  To evaluate the effect of various dose levels of DFV890 versus placebo to reduce circulating levels of inflammatory markers in participants with coronary heart disease and elevated hsCRP

SECONDARY OUTCOMES:
Plasma trough concentrations (Ctrough) of DFV890 at steady state | From Day 22 to End of Study Visit (up to 92 days)
  To assess the pharmacokinetics of DFV890 in participants with coronary heart disease and elevated hsCRP

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (6):
  - Valley Clinical Trials, Northridge, California
  - Excel Medical Clinical Trials LLC, Boca Raton, Florida
  - UF Health Science Center, Jacksonville, Florida
  - Triad Clinical Trials LLC, Greensboro, North Carolina
  - Monument Health Clinical Research, Rapid City, South Dakota
  - Universal Research Group LLC, Tacoma, Washington
- Novartis Investigative Site, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com